CLINICAL TRIAL: NCT02972736
Title: RadiatiOn Dose Among Different EndOvascular Procedures: the RODEO Study
Acronym: RODEO
Status: Completed | Type: Observational
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, MD, PhD, Ospedale Sandro Pertini, Roma
Other Study IDs: Pertini04
Record Dates: First submitted 2016-11-14; First posted 2016-11-23 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Radiation Injuries
Keywords: Radiation dose; percutaneous coronary intervention; Coronary; Interventional radiology; Electrophysiology
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Interventional Cardiology: All procedures performed by interventional cardiologists
  Interventions: Radiation: Radiation dose expressed as DAP
- Electrophysiology: All procedures performed by electrophysiologists
  Interventions: Radiation: Radiation dose expressed as DAP
- Interventional Radiology: All vascular and non vascular procedures performed by interventional radiologists
  Interventions: Radiation: Radiation dose expressed as DAP

INTERVENTIONS:
Radiation: Radiation dose expressed as DAP

SUMMARY:
Retrospective multicenter study aimed to evaluate radiation exposure associated with different interventional procedures involving interventional cardiologists, interventional radiologists and electrophysiologists.

DETAILED DESCRIPTION:
The use fluoroscopically guided interventional procedures is progressively increasing over the past 20 years.Some previous reports have shown that the radiation dose absorbed by interventional cardiologists is the greatest registered by any medical staff exposed to X-rays. However in recent years new procedures have been introduced and validated in the setting of interventional cardiology and radiology and there is wide variation in patient dose among different procedures.

Radiation issue is an important issue for patients and operators due to the acute deterministic effects and most important for the long term stochastic risk of cancer induction: however this problem is often under-evaluated. Even if the stochastic risk is an all-or-none phenomenon for any individual cell, the greater the radiation exposure, the more cells are injured. Moreover non cancerous effects are possible such as cataract formation in the eye and the probability increases with increasing dose.

Radiation dose can be expressed in different ways: the Air Kerma is the amount of energy absorbed in a given mass of air, whereas the Dose Area Product (DAP) is the absorbed dose of radiation across a given surface area. Generally DAP measurements are more accurate than using Air Kerma measurements for the estimation of patient radiation dose as DAP allows for variations in field size. DAP consents a good estimation of the dose to the irradiated tissue and is an indicator for patient cancer risk.

Aim of our study is to evaluate the radiation dose exposure during different fluoroscopically guided interventional procedures comparing different specialties (electrophysiology, interventional radiology, interventional cardiology).

Methods From January 2013 to December 2015 all diagnostic or interventional procedures performed by interventional operators will be included in this multicenter study without exclusion criteria.

Collection of data will be retrospective in a dedicated database. Radiation exposure will be assessed measuring the DAP and fluoroscopy times for each procedure. Moreover for each procedure all the centers are requested to give information about operator, patient and procedure details.

End point of the study The primary end-point of the study is the comparison of DAP dose among interventional cardiologist, electrophysiologist and interventional radiologist procedures.

Secondary end-point of the study is to compare fluoroscopy times among different procedures.

ELIGIBILITY:
Inclusion Criteria:

* All procedures for which DAP values are available

Exclusion Criteria:

* Procedures without DAP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All procedures with DAP data available
Sampling Method: Non-Probability Sample
Enrollment: 17711 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Radiation dose expressed as DAP | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, PhD, Principal Investigator — Ospedale Sandro Pertini - ASL RM2- Rome- Italy